CLINICAL TRIAL: NCT07024927
Title: Complex Arrhythmia Registry（CAR）： Long-term Outcomes of Catheter Ablation for Atrial Fibrillation or Ventricular Tachycardia： A Multicenter， Prospective Cohort Study
Brief Title: Complex Arrhythmia Registry
Acronym: CAR
Status: Not yet recruiting | Type: Observational
Sponsor: Beijing Anzhen Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: KS2025105
Record Dates: First submitted 2025-06-09; First posted 2025-06-17 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Atrial Fibrillation (AF); Ventricular Tachycardia (VT)
Keywords: atrial fibrillation; ventricular tachycardia; ablation; registry study
MeSH Terms: conditions — Atrial Fibrillation; Tachycardia, Ventricular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- PAF: Paroxysmal atrial fibrillation
  Interventions: Procedure: AF ablation
- PeAF: Persistent atrial fibrillation
  Interventions: Procedure: AF ablation
- VT: Ventricular tachycardia
  Interventions: Procedure: VT ablation

INTERVENTIONS:
Procedure: AF ablation — Catheter ablation will be performed under general anesthesia or local anesthesia. Pulmonary vein isolation (PVI) was performed in all patients. Beyond this mandatory step, the specific ablation strategy/protocol and ablation parameters/settings will be determined at the discretion of the operating physicians at each participating center.
  Groups: PAF; PeAF
Procedure: VT ablation — For patients with hemodynamically stable VT, comprehensive chamber mapping (including activation mapping, substrate mapping, and entrainment mapping) is recommended. This aims to elucidate the VT activation sequence and identify the critical isthmus. Precise ablation targeting the isthmus should be performed to terminate the VT. For patients with hemodynamically unstable VT, substrate mapping during sinus rhythm can be performed first. This includes identification of low-voltage zones and abnormal electrograms (e.g., late potentials, local abnormal ventricular activities - LAVAs). Targeted substrate modification ablation should then be conducted based on the mapping findings. For all patients, complete substrate mapping is recommended after VT termination.
  Groups: VT

SUMMARY:
This is a prospective, non-randomized, multicenter observational registry study designed to systematically evaluate the long-term efficacy and safety of catheter ablation for treating atrial fibrillation (AF) and ventricular tachycardia (VT) in Chinese patients.

DETAILED DESCRIPTION:
With the advancement of cardiac electrophysiology, the latest radiofrequency ablation technologies have played a significant role in the treatment of AF and VT. However, long-term outcome data on the application of these advanced techniques in Chinese patients still remains limited. The prospective, non-randomized, multicenter observational registry study will be divided into two cohorts:

1. The AF Cohort will focus on evaluating the effectiveness and safety of different ablation workflows. It aims to redefine the relationship between AF recurrence and long-term outcomes using AF burden, thereby further optimizing treatment strategies for AF.
2. The VT Cohort will primarily assess the application effects of novel technologies in VT treatment.

These data will provide critical reference information for future diagnostic and management strategies for complex arrhythmias.

ELIGIBILITY:
1. Atrial Fibrillation (AF) Cohort:

   * Inclusion Criteria (Patients must meet ALL of the following criteria):

     1. Age ≥ 18 years.
     2. Diagnosed with atrial fibrillation (AF), including paroxysmal AF (PAF) and persistent AF (PsAF).
     3. Scheduled to undergo first-time catheter ablation for AF.
     4. Procedure to be performed using a 3D mapping system.
     5. Provision of signed written informed consent for study participation and willingness and ability to comply with all protocol-required follow-up assessments.
   * Exclusion Criteria (Patients meeting ANY of the following criteria will be excluded):

     1. Severe congenital heart disease (e.g., Tetralogy of Fallot, corrected transposition of the great arteries).
     2. AF secondary to a clearly reversible cause (e.g., hyperthyroidism, post-operative state, acute alcohol intoxication).
     3. Unstable angina pectoris or acute myocardial infarction (MI) within 30 days prior to enrollment/procedure.
     4. Severe active infection (e.g., septic shock, sepsis).
     5. Contraindications to anticoagulation therapy.
     6. Current participation in another interventional clinical trial that may confound the results of this study.
     7. Any other condition where, in the investigator's judgment, the patient is unsuitable for participation in this study.
2. Ventricular Tachycardia (VT) Cohort

   * Inclusion Criteria (Patients must meet ALL of the following criteria):

     1. Age ≥ 18 years.
     2. Diagnosed with ventricular tachycardia (VT) associated with underlying structural heart disease, including:
     3. Ischemic heart disease (e.g., prior MI, coronary artery disease).
     4. Non-ischemic cardiomyopathy (e.g., dilated cardiomyopathy (DCM), arrhythmogenic right ventricular cardiomyopathy (ARVC), hypertrophic cardiomyopathy (HCM)).
     5. Scheduled to undergo first-time catheter ablation for VT.
     6. Procedure to be performed using a 3D mapping system.
     7. Provision of signed written informed consent for study participation and willingness and ability to comply with all protocol-required follow-up assessments.
   * Exclusion Criteria (Patients meeting ANY of the following criteria will be excluded):

     1. VT due to a transient or reversible cause (e.g., acute myocardial ischemia, severe electrolyte imbalance).
     2. Idiopathic ventricular tachycardia (VT occurring in the absence of structural heart disease).
     3. Cardiac surgery within 60 days prior to the planned ablation procedure.
     4. Severe coagulopathy (e.g., platelet count < 50 x 10⁹/L, disseminated intravascular coagulation (DIC)).
     5. Severe heart failure with left ventricular ejection fraction (LVEF) < 20%.
     6. Severe active infection (e.g., septic shock, sepsis).
     7. Current participation in another interventional clinical trial that may confound the results of this study.
     8. Any other condition where, in the investigator's judgment, the patient is unsuitable for participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 4,000 patients who first undergo ablation will be included and divided into three cohorts: 1,000 in the PAF cohort, 2,000 in the PeAF cohort, and 1,000 in the organic VT cohort.
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2031-12 (Estimated); Study Completion 2031-12 (Estimated)

PRIMARY OUTCOMES:
Freedom from any documented atrial arrhythmia in 12 months after the index ablation procedure | From the end of the 3-month blanking period post-ablation to the 12-month follow-up
Composite outcomes of ventricular tachycardia recurrence, cardiovascular hospitalization, or death during the 12-month follow-up | 12 months
  Recurrent ventricular tachycardia is defined as any appropriate implantable cardiac defibrillation therapy (shock or antitachycardia pacing) or documented sustained monomorphic ventricular tachycardia >30 seconds. Cardiovascular rehospitalization is defined as a hospital admission after the randomly assigned procedure for heart failure, procedure-associated complications, or arrhythmic causes during the 12-month follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Deyong Long, Principal Investigator — Beijing Anzhen Hospital
Locations (1):
- Beijing Anzhen Hospital, Capital Medical University, Beijing, China

IPD SHARING:
Plan to Share IPD: No